CLINICAL TRIAL: NCT01585701
Title: A Cancer Research UK Phase I First in Man Study of the Novel AGC Kinase Inhibitor AT13148 Given Orally in Patients With Advanced Solid Tumours.
Brief Title: Phase I Study of AT13148, a Novel AGC Kinase Inhibitor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRUKD/12/001
Record Dates: First submitted 2012-04-25; First posted 2012-04-26 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Advanced Solid Tumours
Keywords: Phase I; Oncology; AGC Kinase inhibitor; Protein Kinase inhibitor; Clinical Trial; Multiple protein kinases
MeSH Terms: conditions — Neoplasms | interventions — AT13148

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: AT13148 — Days 1, 3, 5 of a weekly schedule in dose escalation cohorts of three patients. Continuous dosing until progression or unacceptable toxicity develops up to a maximum of 12 cycles.

SUMMARY:
The purpose of this first clinical study of the noval multiple AGC kinase inhibitor, AT13148, is to identify the recommended dose for future studies in cancer patients by exploring the safety and maximum tolerated dose and biological effects in patients with advanced solid tumours.

DETAILED DESCRIPTION:
AT13148 is a new drug which looks promising in laboratory studies. We now wish to find out if it will be useful in treating patients with cancer. AT13148 is a type of drug called a protein kinase inhibitor. It blocks several different chemical messengers (enzymes) called AGC kinase proteins. These chemical messengers are part of the signaling process within cells which can make cells produce chemicals that trigger and control cell growth and cell death. In some types of cancer these chemical messengers are 'switched on' or 'switched off' permanently due to changes in the genes of cells called "gene mutations" leading to uncontrolled cancer cell growth. AT13148 targets multiple protein kinases from three families of kinases unlike many of the other protein kinase inhibitors currently being tested which target just one or two kinases. This may mean that it will work better and in a wider group of cancer patients. Patients will not be selected to take part based on having these gene mutations for this first trial because we want to learn more about which mutations are most important but this would be the hope for future trials. The patient population anticipated to benefit from this drug includes certain types of breast, prostate and ovarian cancer which more commonly have these gene mutations.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven advanced solid tumours, refractory to conventional treatment, or for which no conventional therapy exists or is declined by the patient. Paraffin-embedded tumour tissue must be available for genetic mutation status testing.
2. Life expectancy of at least 12 weeks
3. World Health Organisation (WHO) performance status of 0, 1 or 2
4. Haematological and biochemical indices within the ranges shown below. These measurements must be performed within 7 days before their first dose of AT13148 taken between Day -7 to -4.

   Laboratory Test Value required

   Haemoglobin (Hb) ≥ 9.0 g/dL

   Absolute neutrophil count ≥ 1.5 x 10^9 /L

   Platelet count ≥ 100 x 10^9/L

   Fasting glucose ≤ 7 mmol/L

   Either:

   Serum bilirubin ≤ 1.5 x upper limit of normal (ULN)

   Or:

   Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x (ULN) unless raised due to tumour in which case up to 5 x ULN is permissible

   Either:

   Calculated creatinine clearance ≥ 50 mL/min

   Or:

   Isotope clearance measurement ≥ 50mL/min (uncorrected)
5. Adequate lung function indicated by a resting oxygen saturation level (on air) ≥ 94%, a CO-transfer factor > 60%
6. 18 years or over
7. Written (signed and dated) informed consent and be capable of co-operating with treatment and follow-up

Exclusion Criteria:

1. Radiotherapy (except for palliative reasons), endocrine therapy (except luteinizing hormone releasing hormone (LHRH) agonists for prostate cancer), immunotherapy or chemotherapy during the previous four weeks (six weeks for nitrosoureas, Mitomycin-C) and 4 weeks for investigational medicinal products) before treatment.
2. Ongoing toxic manifestations of previous treatments. Exceptions to this are alopecia or certain Grade 1 toxicities, which in the opinion of the Investigator and the Drug Development Office (DDO) should not exclude the patient.
3. Symptomatic brain metastases (if present they must have been stable for > 3 months).
4. Ability to become pregnant (or already pregnant or lactating). However, those female patients who have a negative serum or urine pregnancy test before enrolment and agree to use two highly effective forms of contraception (oral, injected or implanted hormonal contraception and condom, have a intra-uterine device and condom, diaphragm with spermicidal gel and condom) during the study and for six months afterwards are considered eligible.
5. Male patients with partners of child-bearing potential (unless they agree to take measures not to father children by using one form of highly effective contraception [condom plus spermicide] during the study and for six months afterwards). Men with pregnant or lactating partners should be advised to use barrier method contraception (e.g. condom plus spermicidal gel) to prevent exposure to the foetus or neonate.
6. Major thoracic or abdominal surgery from which the patient has not yet recovered.
7. At high medical risk because of non-malignant systemic disease including active uncontrolled infection.
8. Known to be serologically positive for Hepatitis B, Hepatitis C or Human Immunodeficiency Virus (HIV).
9. History of auto-immune disease or known allergy to peanuts.
10. Concurrent hypotension defined as a baseline supine blood pressure (BP) systolic < 90 mmHg.
11. Patients receiving anti-hypertensive treatment or treatment with beta- blockers or rate-limiting calcium agents. A washout period of 5 x half- life of the drug should be applied following withdrawal of any of these treatments.
12. Concurrent congestive heart failure, prior history of class III/ IV cardiac disease (New York Heart Association [NYHA]), prior history of cardiac ischaemia or prior history of cardiac arrhythmia. Coronary angioplasty or stenting in the previous 12 months.
13. Patients with a known left ventricular ejection fraction (LVEF) < 50%. A multi-gated acquisition (MUGA) scan or echocardiogram (ECHO) must be performed in all patients.
14. Concurrent diabetes requiring treatment (diet-controlled diabetes would be acceptable).
15. Prior bone marrow transplant or have had extensive radiotherapy to greater than 25% of bone marrow within eight weeks.
16. A history of or underlying interstitial lung disease.
17. Any other condition which in the Investigator's opinion would not make the patient a good candidate for the clinical study.
18. Is a participant or plans to participate in another interventional clinical study whilst taking part in this study. Participation in an observational study would be acceptable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-05; Primary Completion 2018-01-10 (Actual); Study Completion 2018-01-10 (Actual)

PRIMARY OUTCOMES:
Determining a dose at which no more than one patient out of up to six patients at the same dose level experience a highly probably or probably drug-related dose limiting toxicity (DLT).
Determining causality of each adverse event Adverse Event to AT13148 and grading severity according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.02.

SECONDARY OUTCOMES:
Determining the correlation between pharmacokinetic studies and toxicity and/or efficacy.
Any response (stable disease, partial response or complete response) in any of the patients as determined by the Response Evaluation Criteria in Solid Tumours RECIST) criteria version 1.1.criteria version 1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Marsden Hospital, Institute of Cancer Research, Sutton, Surrey, United Kingdom